CLINICAL TRIAL: NCT03278197
Title: Evaluating a Decision Aid in Clinical Practice for Patients With Localized Prostate Cancer
Brief Title: Evaluation of a Web-based Decision Aid Tool for Prostate Cancer Patients
Acronym: ProDecA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other); Zuyderland Medical Centre (Other); VieCuri Medical Centre (Other); Laurentius Ziekenhuis Roermond (Unknown); St.Jans Gasthuis Weert (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-40-19/11-intern-6745
Record Dates: First submitted 2017-02-22; First posted 2017-09-11 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1.Patients (Experimental): Patients diagnosed with prostate cancer and ex-prostate cancer patients:
  * Interviews with patients to define their decisional needs and to determine the barriers and facilitators to the implementation of shared decision making and the decision aid.
  * Navigating through the Treatmentchoice Decisional Tool and think aloud while running the tool
  * Questionnaires
  Interventions: Other: Interviews; Other: Treatmentchoice Decisional Tool; Other: Questionnaires
- 2.Clinicians (Other): Radiotherapy-oncologists, Urologists, General practitioners, Nurses
  * Interviews with patients to define their decisional needs and to determine the barriers and facilitators to the implementation of shared decision making and the decision aid.
  * Navigating through the Treatmentchoice Decisional Tool and think aloud while running the tool
  * Questionnaires
  Interventions: Other: Interviews; Other: Treatmentchoice Decisional Tool; Other: Questionnaires
- 3.Other involved organizations (Other): Patient Organizations and insurance companies Interviews with stakeholders (patients, clinicians, nurses, GP's, patient organizations, insurance companies) to determine the barriers and facilitators to the implementation of shared decision making and the decision aid
  Interventions: Other: Interviews with stakeholders

INTERVENTIONS:
Other: Interviews — Interviews with patients, physicians and general practitioners (GPs) to define patients' decisional needs.
  Arms: 1.Patients; 2.Clinicians
Other: Treatmentchoice Decisional Tool — Patients and physicians navigate through Treatmentchoice Decisional Tool and think aloud while running the tool
  Arms: 1.Patients; 2.Clinicians
Other: Questionnaires — Patients and physicians fill out questionnaires on the usual care, Delphi study
  Arms: 1.Patients; 2.Clinicians
Other: Interviews with stakeholders — Interviews with stakeholders (patients, clinicians, nurses, GP's, patient organizations, insurance companies) to determine the barriers and facilitators to the implementation of shared decision making and the decision aid.
  Arms: 3.Other involved organizations

SUMMARY:
Patients diagnosed with localized prostate cancer may be eligible for different treatment options. MAASTRO Clinic (MAAStricht Radiation Oncology) developed a web-based decision aid tool for these patients. The goal of the tool is to help patients to understand the treatments, and empower the patients to participate in the decision making process. The aim of this study is threefold:

(A) user-testing and validation of the tool, by using a systematically development process compliant with the IPDAS (International Patients Decision Aids Standards) criteria (B) establish the impact of the tool on the decision making process; (C) identify barriers and facilitators for the implementation of shared decision making and the tool in clinical practice.

The study covers 3 phases:

1. Development phase 1.1 Assess decisional needs of patients and clinicians. 1.2 Test patients' and clinicians' comprehensibility, acceptability and usability on the alpha-version of the tool. 1.3 Value clarification: Delphi study with former prostate cancer patients to determine the most important patient preferences and value clarification aspects the decision aid should include.
2. Implementation phase: Develop an implementation and dissemination plan for shared decision-making which is based on the evaluation of barriers and facilitators for the use of patient decision aid tools in clinical practice.
3. Evaluation phase: Establish the impact of on knowledge, decisional conflict and the shared decision-making process, as well as the extent to which clinicians involve patients in decision-making.

A mixed method will be used. It comprises structured interviews combined with think aloud and questionnaires with stakeholders involved in the whole process of development, implementation and evaluation (patients, urologists, radiotherapists, nurses, general practitioners, patient organizations, and insurance companies).

DETAILED DESCRIPTION:
Prostate cancer is the most common malignancy observed among men in industrialized countries, with 1.11 million new cases diagnosed in 2012 . For patients with localized prostate cancer, different treatment options are available; radical prostatectomy, external beam radiotherapy, interstitial radiotherapy also called Brachytherapy (early-stage disease), and 'active surveillance' (low risk patients). The optimal treatment for patients having localized prostate cancer is not unambiguously proven. Different treatment options cause different side effects that may impact the patients' health-related quality of life. The treatment of choice depends on preferences and personal values. In these preference-sensitive choices it is important to involve the patient in the decision-making process. In this process both the practitioner and the patient exchange information and collaborate in the decision, the physician knows more technical information about the disease, the treatment options and the side effects, the patient knows how the treatment options correspond with his lifestyle, values and preferences.

Patient Decision Aids (PDAs) are tools that can help patients to get involved in decision making by clarifying treatment options, outcomes, and personal values. In the development process of a decision aid it is mandatory to follow a systematic and iterative approach to: (a) understand patient's decisional needs; (b) create prototypical tools; (c) evaluate these prototypes with patients and clinicians, and (d) use these results to improve the tool.

Considering the International Patient Decision Aid Standards (http://ipdas.ohri.ca/), the investigators designed an initial prototype, called Treatmentchoice (http://www.treatmentchoice.info). These standards recommend assessing patients and doctors views in decisional needs, use this information to develop an alpha version of the PDA and validate the Treatmentchoice again with patients and doctors to create a beta version.

The aim of this project is user-testing the initial prototype of the Treatmentchoice. This will allow the investigators to follow a systematic development process and to gain knowledge on the validity of approach of the investigators. The project covers 4 activities:

ACTIVITY 1.1: ASSESS DECISIONAL NEEDS: Elicit patients' and clinicians' views on patient's information, expectations, and needs on decision support. Conclusions and recommendations for improvement of Treatmentchoice will be derived and the current prototype will be improved creating an alpha prototype.

ACTIVITY 1.2: ALPHA-TESTING: Testing patients' and clinicians' comprehensibility, acceptability and usability on the alpha prototype. A mixed method will be used; structured interviews combined with think aloud (Ahmed, 2009) and questionnaires (Unified Theory of Acceptance and Use of Technology (UTAUT) - Venkatesh et al.) with both patients and clinicians (urologists, radiotherapists and general practitioners). Conclusions and recommendations will be documented. Considering this assessment, the prototype will be improved. Alpha testing will be repeated with this improved prototype using an iterative process, until the tool is comprehensible, acceptable and usable for both patients and physicians.

ACTIVITY 1.3: DELPHI STUDY: Gain an in-depth understanding of the information needs of prostate cancer patients at each stage from diagnosis to treatment and post-treatment. The purpose is to improve the contents of the decision aid so that it contains an accurate representation of the factors that are most relevant to prostate cancer patients. First, focus group interviews with former prostate cancer patients and patient organizations will be carried out. The results will be analyzed and a list of factors will be generated. A Delphi consensus process will be used to rank the relative importance of these factors and the tool will be updated to give information that is most important for patients.

ACTIVITY 2: IMPACT STUDY (or beta testing): Evaluation of the impact of Treatmentchoice on knowledge, decisional conflict and the shared decision making process, as well as the extent to which clinicians involve patients in decision making. A variety of questionnaires will be used to assess different outcome measures:

* Age and educational level, home internet connection, and computer skills
* Knowledge test will be assessed using 20 statements, which can be rated as "true", "false" or "do not know" .
* Decisional conflict will be assessed using the Decisional Conflict Scale (DCS). This 16-item scale has five subscales: feeling informed, decisional uncertainty, clear values, support, and quality of decisions. Each of these items is scored on a five-point Likert scale from 1 (strongly agree) to 5 (strongly disagree).
* Patient's desire to participate in medical decisions will be assessed using a 5-item Control Preference Scale.
* The Shared Decision Making (SDM) process will be assessed by the perceptions of patients, using the SDM-Q9 instrument for patients. The instrument provides 9 statements, which can be rated on a six-point scale from 0 (completely disagree) to 5 (completely agree). (SDM-Q9, Rodenburg, 2015 /Dutch version).
* The process of SDM will also be assessed by the perceptions of the physician (the urologist or the RTO if the decision is made together with an RTO), using the SDM-Q9 instrument for professionals. The instrument provides 9 statements, also rated on a six-point scale.

The patients will be asked to fill in the questionnaires at two time points: directly after the decision making process and 3 months after the decision making process. Their physician will be asked to fill in the questionnaire at one-time point, directly after the decision making process.

ACTIVITY 3: IMPLEMENTATION: Identify key aspects on the implementation and dissemination for shared decision-making in prostate cancer. Semi-structured interviews will be performed to recognize barriers and facilitators for implementation in clinical practice, to develop strategies for the implementation of decision aids and to facilitate optimal shared decision-making which is tailored to the needs of the end-users (patients and doctors).

ELIGIBILITY:
1. Patients diagnosed with localized prostate cancer. There are no criteria for treatment type.

   * Inclusion criteria:

     * Stage I-II primary prostate cancer
     * Proficient in Dutch
     * > 18 years old
   * Exclusion criteria:

     * Patients that do not have a treatment choice (due to contra-indications or other medical reasons)
     * Patients with recurrent disease.

   For alpha testing patients that already made their decision are selected. For each treatment (external beam radiotherapy (RT), interstitial RT, surgery and active surveillance) at least 10 patients will be included.

   For beta testing patients that are facing their decision will be included. Aiming for an effect size of 0.60 for a difference in mean total score on the Decisional Conflict Scale, it would require 45 patients per group (pre and post intervention) to determine this effect with alpha 0.05 and power 0.80.

   For the Delphi study prostate cancer patients who already underwent treatment will be included.
2. Clinicians:

   * Radiotherapy-oncologists
   * Urologists
   * General practitioners
   * Nurses.

   For alpha testing at least 10 physicians are selected.

   For beta testing at least 45 questionnaires are required.
3. Patient organizations and insurance companies will be interviewed to evaluate barriers and facilitators for implementation in clinical practice. The study will focus on their respective roles in the promotion of shared decision making: patient organizations in raising awareness among patients and insurance companies in providing incentives for the use of decision aids in clinical practice.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Patient's decisional needs to make a decision about their treatment | up to 1 year
  Patients' decisional needs (development phase):semi-structured interviews with patients about their medical history, their experience with the treatment, the decision about their treatment, and what information the patients need to make an informed decision
Comprehensibility of the decision aid too | up to 1 year
  Quantitative research using the Unified Theory of Acceptance and Use of Technology (UTAUT Venkatesh et al. 2013). This questionnaire. (5-Likert) measure how patients and clinicians perceived its utility, effectiveness and efficiency for shared decision-making, as well as their satisfaction with the decision aid.
Usability of the decision aid too | up to 1 year
  Quantitative research using a questionnaire based on the International Standard ISO-9242-11. This questionnaire (5-Likert) measure to what extent the decision aid is easy to use.
Decisional conflict (patients, evaluation phase) | 2 weeks after diagnosis
  Decisional conflict will be assessed using the DCS (Decisional conflict scale): change in DCS between baseline group (usual care) and intervention group (use of the aid tool)
Control Preference Scale (patients; evaluation phase) | 2 weeks after diagnosis
  Patient's preference to participate in medical decisions will be assessed using the 5-item Control Preference Scale (CPS):change in CPS between baseline group (usual care) and intervention group (use of the aid tool)
Perception shared decision-making (patients; evaluation phase) | 2 weeks after diagnosis
  Patient's perception of the shared decision-making process will be assessed using the (shared decision making) SDM-Q9 instrument for patients: change in SDM between baseline group (usual care) and the intervention group (use of the aid tool)
Perception shared decision-making (doctors; evaluation phase) | 2 weeks after diagnosis
  Doctor's perception of the shared decision-making process will be assessed using the SDM-Q9 instrument for professionals: change in SDM between baseline group (usual care) and the intervention group (use of the aid tool)]]

SECONDARY OUTCOMES:
Patients' views on the current decision-making process | upto 1 year
  Patients' views on the current decision-making process (development phase)
Patients' satisfaction with decision aid (Treatmentchoice) | upto 1 year
  Patients' satisfaction with decision aid (Treatmentchoice) (development phase)
Patients' intention to use and recommend Treatmentchoice to others | upto 1 year
  Patients' intention to use and recommend Treatmentchoice to others (development phase)
Insights into the value clarification process of prostate cancer patients | an average of 2 year
  Insights into the value clarification process of prostate cancer patients by questionnaires (development phase)

OTHER OUTCOMES:
Barriers and facilitators for the implementation of Treatmentchoice in clinical practice | an average of 2 years
  Barriers and facilitators for the implementation of Treatmentchoice in clinical practice (implementation phase) will be assessed by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD,PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Maastro Clinic, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No